CLINICAL TRIAL: NCT01314482
Title: The Efficacy of Prophylactic Administration of Minocycline in Reducing Chronic Intercostal Neuralgia Post-thoracotomy
Brief Title: Minocycline for the Prevention of Post-operative Intercostal Neuralgia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Adelaide (Other)
Responsible Party: Principal Investigator, Prof Paul Rolan, Professor of Clinical Pharmacology, University of Adelaide
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U1111-1119-6985
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Post-operative Intercostal Neuralgia
Keywords: Neuropathic pain; Minocycline
MeSH Terms: conditions — Neuralgia; cyclopia sequence | interventions — Minocycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Minocycline (Experimental)
  Interventions: Drug: Minocycline

INTERVENTIONS:
Drug: Minocycline — 200mg bd for 3 days before surgery

SUMMARY:
In about half the patients who have an open chest surgery there is persistent severe pain in the chest. The investigators are examining whether minocycline, a commonly used antibiotic, will prevent pain. Minocycline blocks the activity of immune cells which the investigators believe are responsible for prolonging the pain.

DETAILED DESCRIPTION:
The study is of double-blind placebo controlled parallel groups design in up to 116 patients undergoing elective open thoracotomy. Minocycline 200mg twice daily or matching placebo are given three days before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Aged 18 years or older
* Undertaking elective, open thoracotomy with ample time pre-operatively to provide informed consent and undertake dosing
* Sufficient fluency in English language to read and understand consent form, fulfil study requirements and communicate with research staff
* Negative pregnancy test at screening for women of child bearing potential
* Females of child bearing potential must agree to use a medically acceptable method of contraception other than oral contraceptives from time of first dosing until one week post-operatively. Acceptable methods include abstinence, contraceptive patches, NuvaRing (etonogestrel/ethinyl oestradiol vaginal ring), diaphragm with vaginal spermicide, intrauterine device, condom and vaginal spermicide, progestin implant or injection
* Avoid prolonged, direct sunlight or ultra-violet light exposure during dosing period
* Refrain from strenuous activities and avoid changes to regular exercise patterns throughout trial period

Exclusion Criteria:

* Pregnant or breast feeding
* Known allergy to minocycline and other tetracycline antibiotics
* Pre-existing neuralgic pain condition in area designated for operation
* Physical abnormality in area designated for operation
* Taking disallowed concomitant medication
* Renal insufficiency as determined by a calculated creatinine clearance of < 60mL/min
* Hepatic dysfunction as determined by alanine transaminase and/or aspartate transaminase in excess of three times upper normal limits
* Diagnosis of systemic lupus erythematosus
* Recent diagnosis of enterocolitis or colitis
* Participation in another trial of an investigational product within 30 days of commencing dosing or are scheduled to commence trial of an investigational product during study period
* Patients who, in an Investigator's opinion, should not participate in the trial or may not be capable of following the trial schedule for any reason
* History of major psychiatric disorder not medically controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Daily pain scores on a numerical rating scale | 3 months

SECONDARY OUTCOMES:
Hypo/hyperaesthesia to punctate sensation | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia